CLINICAL TRIAL: NCT03248453
Title: Do Feedback Given by an Automatic and Objective System in Simulated Colonoscopy Increase Learning and Time Spent Practicing? A Randomized Trial
Brief Title: Feedback Given by an Automatic and Objective System in Simulated Colonoscopy Increase Learning and Time Spent Practicing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Andreas Slot Vilmann, MD. Andreas Slot Vilmann, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COPS/self-regulated feedback
Record Dates: First submitted 2016-10-13; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Simulation Training; Education, Medical
Keywords: Simulated colonoscopy; Self-regulated learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoPS feedback (Experimental): Each participant will as feedback be given the actual CoPS after reaching the cecum on the standardized Kagaku Training Model. A leaderboard with experts performances will be present for comparison.
  Interventions: Other: CoPS
- No CoPS feedback (No Intervention): No feedback is given and the participants are not aware of the CoPS

INTERVENTIONS:
Other: CoPS — The COPS is an automated and objective computer-based program which generate a score/number after the colonoscope has reached the cecum. The participants are able to compare the score with experts.
  Arms: CoPS feedback

SUMMARY:
The aim is to investigate if feedback given by an automatic and objective system in simulated colonoscopy (the investigation of the large intestine) increase learning and time spent practicing.

DETAILED DESCRIPTION:
A standardized Kagaku Colonoscopy Training Model (Kyoto Kagaku Co Ltd, Kyoto, Japan) in combination with an Olympus colonoscope, a monitor and a Magnetic Endoscope Imaging (MEI) Scope Guide (Olympus Medical systems Corp) is used. The Kyoto Kagaku Colonoscope Training Model is a phantom model in full-size of the human colon. The model consists of an abdomen model, a soft and flexible rubber colon, anal sphincter opening and an abdomen skin cover. The rubber colon provides a realistic life-like response, which makes the participants able to feel when the colonoscope stretch and bent the rubber colon. To reduce friction between the rubber colon and the colonoscope a lubricant gels is applied inside the rubber colon. By hand pump the anal sphincter is manipulated, allowing insufflation and suction. Six different cases with different level of difficulty are possible. We chose case 2 (simple layout, but a long sigmoid colon) and case 4 (a challenging layout, with a difficult-to-shorten sigmoid colon and a drooping transverse colon) for training cases. Case 3 (simple layout, but with a naturally formed "Alpha" loop in the sigmoid colon) is chosen for the final test.

Experts - 10 experts, defined by the number of colonoscopies in total (> 1000), colonoscopies done within the last year (> 150) and locally considered among the best, will be recruited voluntarily. The experts are introduced to the Colonoscopy Training Model and allowed 15 minutes of practices before tests is recorded. With the exception of the first expert who is given the best Colonoscopy Progression Score (CoPS) executed by an instructor, the experts are shown the other experts top scores for each case as a motivation. Each expert carries out three different cases: Case 2, 3 and 4. Time for each case are 15 minutes.

Novices - 44 novices (interns and junior residents) with no experience in colonoscopy will be enrolled through a volunteer application form in the study. All novices will be handed written information about colonoscopy in general and basics. Novices will be introduced to the technical characteristics of the colonoscope by an instructor and allowed training for 15 minutes before the data collection is started. No feedback (from instructors) will be given during the training. Instructors will start data collection with introduction of the colonoscope into the anus and the data collection is stopped when the cecum is reached. For training the novices will have a free choice between case 2 and 4. Each novice is given the opportunity to redo the training for as long as they like before they believe to be ready for the final case. Case 3 will be used for the final test and all participants are to complete the case tree times.

Novices will be randomized into two groups:

1. The intervention group is given feedback; presented with the CoPS after each time they reach cecum. A leaderboard, presenting all the experts CoPS, for comparison and motivation will be present next to the phantom model.
2. Control group is not given any CoPS.

ELIGIBILITY:
Inclusion Criteria:

* Physicians
* No endoscopic experience

Exclusion Criteria:

* Non-physicians
* Previous experience with endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Final CoPS | There is only one time point (baseline = after the final cases)
  The final CoPS is a mean-score of the CoPS´ in the final cases. Primary outcome is the difference between the interventiongroup and the control group.

SECONDARY OUTCOMES:
Total time spent practicing | up to 120 minutes
  Difference in total time spent practicing between groups
Amount of time spend on each case | up to 720 seconds
  Time spent practicing on case 2 versus time spent practicing on case 4

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, Professor, Principal Investigator — CAMES-Rigshospitalet, Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Acedemy of Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaltenbach T, Leung C, Wu K, Yan K, Friedland S, Soetikno R. Use of the colonoscope training model with the colonoscope 3D imaging probe improved trainee colonoscopy performance: a pilot study. Dig Dis Sci. 2011 May;56(5):1496-502. doi: 10.1007/s10620-011-1614-1. Epub 2011 Mar 16. PMID 21409379
- [Background] Nerup N, Preisler L, Svendsen MB, Svendsen LB, Konge L. Assessment of colonoscopy by use of magnetic endoscopic imaging: design and validation of an automated tool. Gastrointest Endosc. 2015 Mar;81(3):548-54. doi: 10.1016/j.gie.2014.07.019. Epub 2014 Sep 23. PMID 25257129
- [Background] Plooy AM, Hill A, Horswill MS, Cresp AS, Watson MO, Ooi SY, Riek S, Wallis GM, Burgess-Limerick R, Hewett DG. Construct validation of a physical model colonoscopy simulator. Gastrointest Endosc. 2012 Jul;76(1):144-50. doi: 10.1016/j.gie.2012.03.246. PMID 22726473
- [Background] Brinkman WM, Buzink SN, Alevizos L, de Hingh IH, Jakimowicz JJ. Criterion-based laparoscopic training reduces total training time. Surg Endosc. 2012 Apr;26(4):1095-101. doi: 10.1007/s00464-011-2005-6. Epub 2011 Nov 1. PMID 22042592
- [Background] Strandbygaard J, Bjerrum F, Maagaard M, Winkel P, Larsen CR, Ringsted C, Gluud C, Grantcharov T, Ottesen B, Sorensen JL. Instructor feedback versus no instructor feedback on performance in a laparoscopic virtual reality simulator: a randomized trial. Ann Surg. 2013 May;257(5):839-44. doi: 10.1097/SLA.0b013e31827eee6e. PMID 23295321
- [Background] Wulf G, Raupach M, Pfeiffer F. Self-controlled observational practice enhances learning. Res Q Exerc Sport. 2005 Mar;76(1):107-11. doi: 10.1080/02701367.2005.10599266. No abstract available. PMID 15810775
- [Background] Park HJ, Hong JH, Kim HS, Kim BR, Park SY, Jo KW, Kim JW. Predictive factors affecting cecal intubation failure in colonoscopy trainees. BMC Med Educ. 2013 Jan 19;13:5. doi: 10.1186/1472-6920-13-5. PMID 23331720
- [Derived] Vilmann AS, Norsk D, Svendsen MBS, Reinhold R, Svendsen LB, Park YS, Konge L. Computerized feedback during colonoscopy training leads to improved performance: a randomized trial. Gastrointest Endosc. 2018 Nov;88(5):869-876. doi: 10.1016/j.gie.2018.07.008. Epub 2018 Jul 19. PMID 30031803